CLINICAL TRIAL: NCT03475823
Title: The Acute and Chronic Cognitive and Cerebral Blood Flow Effects of a Sideritis Scardica (Mountain Tea) Extract: a Double Blind, Randomized, Placebo Controlled, Parallel Groups Study in Healthy Humans
Brief Title: Cognitive and Blood Flow Effects of Mountain Tea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Finzelberg (Unknown)
Responsible Party: Principal Investigator, Emma Wightman, Principal investigator, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SUB010_Khan_141116
Record Dates: First submitted 2018-02-15; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Cognitive Change; Affect; Blood Pressure; Neuroimaging
MeSH Terms: interventions — Ginkgo Extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All treatment was prepared and randmised by a third-party researcher who had no further involvement in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo control (Placebo Comparator): Inert comparator indistinguishable from active interventions
  Interventions: Dietary Supplement: Placebo control
- Active control (Active Comparator): 240 mg ginkgo biloba
  Interventions: Dietary Supplement: Ginkgo biloba
- Low dose sideritis scardica (Experimental): 475 mg sideritis scardica
  Interventions: Dietary Supplement: Sideritis Scardica
- High dose sideritis scardica (Experimental): 950 mg sideritis scardica
  Interventions: Dietary Supplement: Sideritis Scardica

INTERVENTIONS:
Dietary Supplement: Sideritis Scardica — Sideritis Scardica is a popular, naturally un-caffeinated Eastern European tea extract derived from the ironwort plant
  Other Names: Shepherd's tea; Olympus tea; Mountain tea
  Arms: High dose sideritis scardica; Low dose sideritis scardica
Dietary Supplement: Ginkgo biloba — Ginkgo biloba is an extract from the ginkgo tree comprising ginkgolides and bilobalide. In this trial Ginkgo acted as an active control.
  Arms: Active control
Dietary Supplement: Placebo control — An inert encapsulated powder provided by Finzelberg.
  Arms: Placebo control

SUMMARY:
Two doses (475 mg and 950 mg) of Sideritis Scardica (SS or 'mountain tea') are investigated for cognitive, mood, blood pressure and cerebral blood flow effects in a healthy group of 50-70 yr olds, both acutely and following 28 days of consumption.

DETAILED DESCRIPTION:
The presence of polyphenols such as ferulic acid, chlorogenic acid and apigenin in Sideritis Scardica (SS or 'mountain tea') are likely responsible for the cognitive and mood effects of its consumption and this could be underpinned by the ability of such polyphenols to prevent monoamine neurotransmitter reuptake and to increase cerebral blood flow (CBF).

The current randomised, placebo controlled, parallel groups study extends on the abovementioned small amount of literature; assessing both cognitive and mood outcomes in a sample of older (50-70 yrs) adults, as well as blood pressure (BP) and CBF, in a sub-sample, utilizing near-infrared spectroscopy (NIRS). The above will be assessed acutely (pre-dose and 90- and 310-mins post dose) on day 1 and following 28 days consumption of either a placebo control, and active control of 240 mg ginkgo biloba, 475 mg SS or 950 mg SS.

ELIGIBILITY:
Inclusion Criteria:

* 50-70 yrs of age
* No underlying health problem which would prevent engagement with the study

Exclusion Criteria:

* BMI < 18 or > 35 kg/m2
* High blood pressure (defined as systolic > 159 mmHg or diastolic > 90 mmHg)
* Smoking
* Food allergies or insensitivities
* Pregnancy or breast feeding
* Currently taking any medication (use of contraceptives/hormone replacements was not excluded) or dietary supplements which would contraindicate with the study
* Sleep disturbances and/or taking sleep aid medication
* History of neurological, vascular or psychiatric illness
* Current diagnosis of anxiety or depression
* Migraines
* Recent history (within 12 months) of alcohol/substance abuse
* Disorder of the blood
* Heart disorder/history of vascular illness
* Respiratory disorder requiring regular medication
* Type I or II diabetes
* Renal disease, hepatic disease or severe disease of the gastrointestinal tract - Any health condition that would prevent the fulfilment of the study requirements

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Changes in cognition | Pre-dose and 90- and 310-mins post-dose on day 1 and on day 28 of consumption
  Acute and chronic change in cognitive function via the following cognitive tasks: numeric working memory, choice reaction time, corsi blocks, serial 3 and 7 subtractions, rapid visual information processing, peg and ball, name to face recall, picture recognition, word recognition, immediate word recall and delayed word recall. All tasks provide an outcome for accuracy, speed and error.

SECONDARY OUTCOMES:
Cerebral Blood Flow | Pre-dose and between ~150-240-mins post-dose on day 1 and on day 28 of consumption
  Blood flow changes measured in the pre-frontal cortex utilizing Near-Infrared Spectroscopy (NIRS). Outcome measures include; oxygen saturation, oxygenated haemoglobin, deoxygenated haemoglobin and total haemoglobin.
Changes in mood | On day 1 and following 28 days of consumption
  Acute and chronic changes in mood as assessed by the State-Trait anxiety Inventory (Spielberger, 1983) and Bond-Lader (1974) visual analogue scales. For both measures a baseline score is calculated and all subsequent post-dose scores are subtracted from this to produce change (change from baseline) scores. Both the STAI and Bond-Lader scales produce numerical values and the outcome measure for both will be the same; i.e. changes in this numerical value from baseline mood.
Blood Pressure | Pre-dose and 90- and 310-mins post-dose on day 1 and on day 28 of consumption
  Acute and chronic changes in blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Emma L Wightman, PhD, Principal Investigator — Northumbria University
Locations (1):
- Brain Performance and Nutrition Research centre, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided